CLINICAL TRIAL: NCT01348152
Title: A Randomized, Double-Blinded, Placebo-Controlled Exploratory Study of Daikenchuto (TU-100) in Patients With Functional Constipation
Brief Title: Effect of TU-100 in Patients With Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TU100CPT3
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Functional Constipation
Keywords: Gastric Emptying
MeSH Terms: interventions — dai-kenchu-to; 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo TID
  Interventions: Drug: Placebo
- DAIKENCHUTO (TU-100) 15 g/day (Experimental): TU-100 5g TID
  Interventions: Drug: DAIKENCHUTO (TU-100)

INTERVENTIONS:
Drug: DAIKENCHUTO (TU-100) — Subjects will be randomized to 15 g/day of TU-100. Dosage is granule. Subjects will ingest two 2.5 g doses of TU-100 three times daily for 34 consecutive days.
  Arms: DAIKENCHUTO (TU-100) 15 g/day
Drug: Placebo — Subjects will be randomized to 15 g/day of placebo. Dosage is granule. Subjects will ingest two 2.5 g doses of placebo three times daily for 34 consecutive days.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the improvement in the severity of constipation (from Baseline to Day 28), determined by the constipation severity instrument (CSI) score [1], compared to placebo, following a total daily oral dose of 15 g TU-100 administered for 28 consecutive days in adult subjects with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Have severity of constipation in CSI score of 25 to 74 points.
2. Have the ability to orally ingest study medication, TU-100, and the SmartPill capsule.
3. Be male or female aged between 18 and 80 years old, inclusive.
4. Provide written informed consent before participation in the study after full explanations of the study purpose and procedures.
5. If a female is of childbearing potential and sexually active:

   1. She must agree to practice a highly effective method of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, during their participation in the trial and for 4 weeks after receiving the last dose of study drug
   2. She must have a negative serum pregnancy test before randomization.
6. If a male is sexually active with a female of childbearing potential:

   1. He must agree to use a double barrier of birth control during the study and for 4 weeks after receiving the last dose of study drug.
   2. He must not donate sperm during the study and for 4 weeks after receiving the last dose of study drug.

Exclusion Criteria:

1. Presence of strictures, fistulas, or physiological or mechanical bowel obstruction.
2. Presence of implanted or portable electro-mechanical medical devices.
3. History of gastric bezoar or swallowing disorders.
4. History of gastrointestinal surgery within 3 months of screening.
5. History of bowel resection.
6. Current pregnancy or lactation.
7. History of clinically significant alcohol or drug abuse within a year of screening.
8. Have any other condition that might adversely affect capacity to participate in this study, including liver disorders (with serum alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] levels exceeding 2.5 times the upper limit of normal [ULN]), kidney disorders, heart failure, blood disorders, or metabolic disorders.
9. Be diagnosed with cancer, ulcerative colitis, Crohn's disease, diverticulitis, scleroderma, Hirschsprung's disease, Chagas' disease, multiple sclerosis, Parkinson's disease, stroke, paraplegia, quadriplegia, insulin-dependent diabetes mellitus, untreated hypothyroidism, or any other systemic or psychiatric disorder which may, in the opinion of the investigator, interfere with the evaluation of TU-100.
10. Be taking any medication as follows: anticholinergic agents/medications with anticholinergic effect (list of prohibited drugs attached in Appendix G; antidepressants are permissible if the patient's symptoms are stable, and the doses are NOT changed during the course of the study), warfarin, prokinetics (i.e., Domperidone, Metoclopramide), narcotic analgesics, or any agent that might interfere with the evaluation of TU-100 in the opinion of the investigator.
11. Have a history of allergic reaction or hypersensitivity to ginseng, ginger, and Sichuan pepper.
12. Have severe dysphagia to food or pills.
13. Have participated in any other clinical study within 30 days before enrolling in this study.
14. Be unsuitable for participation in this trial for any reason, according to the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Day 28 in CSI total score | Up to 10 weeks

SECONDARY OUTCOMES:
Change from baseline in GI transit time measured by SmartPill capsule. | Up to 10 weeks
Change from baseline to Day 28 in CRQOL total score. | Up to 10 weeks
Changes from baseline in stool frequency, stool consistency, severity of straining, and completeness of evacuation determined from entries in the bowel pattern diary. | Up to 10 weeks
Change from baseline to Day 28 in CSI subscale scores. | Up to 10 weeks
Change from baseline to Day 28 in CRQOL subscale scores. | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anders F Mellgren, MD, PhD, Principal Investigator — Colon and Rectal Surgery Associates
Locations (1):
- Colon and Rectal Surgery Associates, Minneapolis, Minnesota, United States